CLINICAL TRIAL: NCT02361164
Title: Prospective Two-year Observational Study to Evaluate the Effect of Bacterial Colonisation of the Nasopharynx on the Occurence of Acute Respiratory Infections in a Birth Cohort of Children and Their Mothers
Brief Title: Birth Cohort Study for Respiratory Infections
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.11.NRC
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, clinical samples for bacterial and viral isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mother/child pair: Mother/child pair.

SUMMARY:
The primary objectives are to evaluate relationship between nasopharyngeal microbial colonization and the occurrence of AOM or pneumonia in infants.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Parity: any but with history of previous normal delivery
* Weight: Body Mass Index greater than 18.5 but less than 35
* Past obstetric history: Uncomplicated pregnancy, unremarkable medical and obstetric conditions
* Current pregnancy: Uneventful progression of pregnancy
* General health: Normal health related functional status during pregnancy
* Singleton pregnancy as determined by clinical examination and/or by ultrasonography
* Cephalic presentation as determined by abdominal clinical examination
* Expected to have normal pregnancy related outcome
* Written informed consent

Exclusion Criteria:

* Medical history: Known history of diabetes, hypertension, or any systemic disorder
* Gynecological history: History of major gynecological problem/treatment
* Complications in previous pregnancy
* Previous obstetric cholestasis
* Previous acute fatty liver disease
* Conditions during current pregnancy

  1. RhD negative mother
  2. APH/Placental abruption
  3. Placenta Praevia
  4. Unstable lie
  5. Multiple pregnancy
  6. Pregnancy induced hypertension (systolic > 140 mm of Hg, diastolic > 90 mm of Hg)
  7. Severe pre-eclampsia or eclampsia
  8. Gestational diabetes
  9. Onstetric cholestasis
  10. Current history of drug/alcohol abuse
  11. BMI of less than 18.5 or more than 35. Severe pallor as detected clinically or by HB level (< 7 gm/dL), and oedema
  12. Blood samples drawn and tested for VDRL (Positive VDRL) Cephalopelvic disproportion (CPD)
  13. History of taking antibiotic within 3 weeks prior to this study
  14. Patient unwilling to comply with study protocol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory disease (Acute Otitis Media, Acute Respiratory Infection) | 2 years
Naso-/oro-Pharyngeal colonization with specific pathogens and microbiota | 2 years
Risk factors for recurrent Upper Respiratory Track Infection in terms of bacteria or virus, nutritional and immune status, as well as epidemiological factors | 2 years

SECONDARY OUTCOMES:
Incidence of maternal urogenital infection | 2 years
Birth outcome | 2 years

OTHER OUTCOMES:
Evaluation of FUT2/3 polymorphism and association with infant health outcomes | One time point during the study
  Analysis on saliva samples
Incidence of diarrhea and evaluation of gut health in infants | 2 years
  Analysis of fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Shafiqul Alam Sarker, M.D., Principal Investigator — International Center for Diarrheal Disease Research, Bangladesh
Locations (1):
- International Center for Diarrheal Disease Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No